CLINICAL TRIAL: NCT03553355
Title: Effects of Infrared Laser Moxibustion on Cancer-related Fatigue in Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 81603703
Record Dates: First submitted 2018-05-04; First posted 2018-06-12 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Cancer-related Fatigue
Keywords: infrared laser moxibustion; cancer-related fatigue; breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Infrared Laser Moxibustion Therapy (Experimental): Each patient will receive this treatment twice per week for six weeks (12 sessions total).
  Interventions: Device: Infrared Laser Moxibustion
- Sham Infrared Laser Moxibustion Therapy (Sham Comparator): The patients will receive treatment from sham laser moxibustion instrument.
  Interventions: Device: Sham Infrared Laser Moxibustion
- Waitlist Controls (No Intervention): The patients maintain their usual treatment and self-care,

INTERVENTIONS:
Device: Infrared Laser Moxibustion — We will use SX10-C1 laser moxibustion devices (Shanghai Wonderful Opto-Electrics Tech Co Ltd, Shanghai, China) for the ILM and SILM groups. Four laser probes will be synchronously aligned with 4 points (tST36 (bilateral), CV4, and CV6 acupoints) and we will irradiate each acupoint 2 cm away from the skin surface for 20 minutes. Each patient will receive this treatment twice per week for six weeks (12 sessions total).
  Arms: Infrared Laser Moxibustion Therapy
Device: Sham Infrared Laser Moxibustion — The sham laser moxibustion instrument appears to be identical as the real one.
  Arms: Sham Infrared Laser Moxibustion Therapy

SUMMARY:
Cancer-related fatigue (CRF) is the most common and distressing symptom associated with tumor or cancer treatment that breast cancer survivors (BCS) experience.The investigators previously found the laser moxibustion was potentially efficacious for CRF; however, more rigorously designed study is needed to confirm its benefit. The primary aim of this study is to determine the efficacy of 10.6µm infrared laser moxibustion and its long-term effects on CRF. Secondary aims are to evaluate the effect of infrared laser moxibustion on co-existing symptoms such as among BCS experiencing CRF.

DETAILED DESCRIPTION:
The randomized, placebo-controlled, three-arm trial will be conducted to evaluate the efficacy of infrared laser moxibustion (ILM) and sham ILM (SILM) compared to waitlist control (WLC) for moderately to severely fatigued BCS. The two intervention groups will receive real/sham infrared laser moxibustion on four acupoints (e.g. ST36 (bilateral), CV4, and CV6) for 20 minutes each session for six weeks (two times per week). The primary endpoint is the change in fatigue scores from Baseline to Week 6 as measured by the Chinese version of the Brief Fatigue Inventory (BFI-C). Our secondary aims are to compare the severity of comorbidities (e.g. depression, insomnia, and pain) and biological outcomes (e.g. telomere length) among the three groups.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 years and 75 years
* Breast cancer survivors with a diagnosis of stage I-IIIa
* Cessation of cancer-related treatments (e.g. surgery, chemotherapy, radiotherapy) at least 12 weeks before the trial, with the exception of hormonal and trastuzumab therapy
* Complaint of fatigue starting on or after their cancer diagnosis,Brief Fatigue Inventory score of ≥ 4

Exclusion Criteria:

* Severe anemia (platelet count <60,000/μL,hemoglobin <8 g/dL, or leukocyte count<3000/μL)
* Abnormal findings in a thyroid function test (abnormal level of free thyroxine and thyroid stimulating hormone <0.1 μIU/ml or TSH> 5.1 μIU/ml)
* Having received acupuncture for any indication in the previous 4 weeks or having received acupuncture test within the past 6 months.
* Untreated major depressive disorder and suicidal ideations.
* Pregnant or planning to become pregnant

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2021-03-23 (Actual); Study Completion 2021-07-27 (Actual)

PRIMARY OUTCOMES:
Chinese version of the Brief Fatigue Inventory (BFI-C) | Change from Baseline BFI-C at 6 weeks
  The Chinese version of the Brief Fatigue Inventory (BFI) : It uses 10-point numeric descriptions: scores of 1 to 3 represent mild levels of fatigue, scores of 4 to 6 represent moderate levels of fatigue, and scores of 7 to 10 represent severe levels of fatigue.

SECONDARY OUTCOMES:
Quality of Life (QOL) | 0week; 3weeks；6weeks; 12weeks; 18weeks
  The Chinese version of the Functional Assessment of Cancer Therapy-Breast (FACT-B) : It is a 37-item instrument and each question is rated on a 5-point Likert scale. Higher scores represent improved global quality of life.
Depression/Anxiety | 0week; 3weeks；6weeks; 12weeks; 18weeks
  The Chinese version of the Hospital Anxiety and Depression Scale (HADS): The HADS is a brief 14-item instrument, with seven items in each of the anxiety and depression scales that are scored from 0 to 3, resulting in scale scores that range from 0 to 21 Established cutoffs are: 0-7 not significant, 8-10 subclinical, and 11-21 clinically significant depression/anxiety.
Stress | 0week; 3weeks；6weeks; 12weeks; 18weeks
  The Chinese version of 10-Item Perceived Stress Scale (PSS-10) : It is a 10-item instrument and each question is rated on a 5-point Likert scale (0 = never to 4 = very often). A higher score indicates greater stress.
Insomnia | 0week; 3weeks；6weeks; 12weeks; 18weeks
  The Chinese version of the Pittsburgh Sleep Quality Index (PSQI) : It is a 19-item self-report instrument that includes 7 component scores. The scores for these components range from 0 (no difficulty) to 3 (severe difficulty) and a higher score denoting poorer sleep quality (range: 0-21). It suggested a cut-off of the global score at ⩾8 for the presence of sleep disturbance in cancer patients.
Brief Pain Inventory | 0week; 3weeks；6weeks; 12weeks; 18weeks
  Chinese version of the Brief Pain Inventory (BPI)：It is a 11-item self-administered questionnaire that includes two main scores: a pain severity score (scored from 0 to 10, range from 0 to 40) and a pain interference score (scored from 0 to 10, range from 0 to 70). Higher scores represent worse pain.
Treatment Expectancy | 0week; 3weeks；6weeks
  Acupuncture Expectancy Scale (AES)：It is a 4-item instrument designed to assess outcome expectancy in acupuncture clinical trials, each with a 5-point Likert scale ranging from 1 to 5. The scores range between 4 and 20, with a higher score indicating greater expectancy.

CONTACTS AND LOCATIONS:
Overall Officials: Huijuan Mao, MD, Principal Investigator — Shanghai University of TCM
Locations (1):
- Yueyang Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mao H, Mao JJ, Chen J, Li Q, Chen X, Shen X, Zhao L, Wei J, Shen X. Effects of infrared laser moxibustion on cancer-related fatigue in breast cancer survivors: Study protocol for a randomized controlled trial. Medicine (Baltimore). 2019 Aug;98(34):e16882. doi: 10.1097/MD.0000000000016882. PMID 31441863